CLINICAL TRIAL: NCT05701033
Title: Does Engagement with Heritage Sites Have the Potential to Improve Sub-clinical Levels of Low Wellbeing in NHS Staff: a Feasibility Study. the HerWellNHS Study
Acronym: HerWellNHS
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: PHU/2022/68
Record Dates: First submitted 2022-12-13; First posted 2023-01-27 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Access to heritage — Unmediated access to heritage sites for wellbeing

SUMMARY:
This feasibility study will focus on assessing and identifying the wellbeing effects of self-directed (unmediated) visits to heritage sites for a high-risk population, specifically NHS staff at PHU self-reporting sub-clinical levels of low wellbeing. In particular, it seeks to understand whether wellbeing effects can be derived from unmediated visits to heritage sites, how much exposure to heritage is necessary to experience wellbeing effects, whether and how benefits may be accumulated, how long wellbeing effects may last following visits, and the nature of these wellbeing effects. In addition, it will establish appropriate psychological measures (qualitative and quantitative), test a web-based data collection interface, examine participant choices and their characteristics, and assess participant adherence and response rates prior to developing a clinical trial.

DETAILED DESCRIPTION:
This feasibility study will use quantitative and qualitative psychological measures to examine participant choices of heritage sites and their characteristics, as well as assessing participant adherence and response rates prior to development of a future clinical trial.

It will act as proof of concept, generating a case for the promise of unmediated heritage visits as an effective mental health intervention.

The project will focus on assessing and identifying the wellbeing effects of unmediated visits to heritage sites for NHS staff, and seeks to understand how much exposure to heritage is necessary to experience wellbeing effects, how benefits may be accumulated, how long wellbeing effects may last following a visit, and what the nature of these wellbeing effects may be. The study also seeks to capture the staff experience of engaging with heritage sites, what are the aspects which might result in positive change as a result of the interactions as well if there are any potential risks associated with such interventions.

This project is funded by Historic England. The project partners are as follows: Portsmouth University NHS Hospitals, The Royal Navy National Museum, The Mary Rose Museum, Wessex Archaeology, Portsmouth City Council, Art as Media and the University of Southampton.

ELIGIBILITY:
Inclusion Criteria:

The participant must meet ALL of the following criteria to be considered eligible for the study:

* Male or Female, aged 18 years or above.
* Self-reported subclinical levels of low wellbeing
* Participant is willing and able to give informed consent for participation in the study.
* NHS Staff at Portsmouth Hospitals University NHS Trust

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Having been diagnosed with and/or received treatment for any mental health issues in the past 12 months
* Under 18
* Unable to give informed consent for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Portsmouth Hospitals University NHS Trust staff with self-reported sub-optimal levels of wellbeing
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
improve sub-clinical levels of low wellbeing for staff | Through study completion, an average of 6 months
  As a primary objective, this feasibility study aims to determine whether engagement with heritage sites has the potential to improve sub-clinical levels of low wellbeing for staff at Portsmouth Hospitals University NHS Trust.

SECONDARY OUTCOMES:
What intensity of exposure to heritage is necessary to experience wellbeing effects, and whether and how benefits may be accumulated? | Through study completion, an average of 6 months
  What intensity of exposure to heritage is necessary to experience wellbeing effects, and whether and how benefits may be accumulated?
What kinds of wellbeing benefits do staff experience? | Through study completion, an average of 6 months
  What kinds of wellbeing benefits do staff experience?
What other 'spin-off' effects might be obtained through improved staff wellbeing via visits to heritage sites? | Through study completion, an average of 6 months
  What other 'spin-off' effects might be obtained through improved staff wellbeing via visits to heritage sites?
What factors are related to the wellbeing effects of heritage visits (e.g. exercise, being with other people, duration of visit, type of heritage visit)? | Through study completion, an average of 6 months
  What factors are related to the wellbeing effects of heritage visits (e.g. exercise, being with other people, duration of visit, type of heritage visit)?
What is the duration of post-visits effectiveness on wellbeing? | Through study completion, an average of 6 months
  What is the duration of post-visits effectiveness on wellbeing?

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals University NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data to be pseudo anonymised where possible and only available to thre research team